CLINICAL TRIAL: NCT00724659
Title: An Evaluation of Pre and Post Arthrogram Ultrasound Images of Joints: Does Arthrography Have a Role in Ultrasonography?
Brief Title: Pre and Post Arthrogram Ultrasound Images of Joints
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jon Jacobson, Principal Investigator, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2004-0761
Record Dates: First submitted 2008-07-28; First posted 2008-07-29 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Joint Abnormalities
Keywords: Arthrogram; Contrast; Joint; Ultrasound
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound Pre-Arthrogram (Experimental): Ultrasound of the joint(s) before the clinically scheduled arthrogram of the same joint(s)
  Interventions: Procedure: Ultrasound
- Ultrasound Post-Arthrogram (Experimental): Ultrasound of the joint(s) after the clinically scheduled arthrogram of the same joint(s), performed while the body still has a contrast agent in it from the arthrogram. The contrast agent varies with different joint areas, but is usually iodine based (like Ultravist.)
  Interventions: Procedure: Ultrasound

INTERVENTIONS:
Procedure: Ultrasound — Ultrasound of the joint(s) before the clinically scheduled arthrogram of the same joint(s)
  Arms: Ultrasound Pre-Arthrogram
Procedure: Ultrasound — Ultrasound of the joint(s) after a clinically scheduled arthrogram is performed. Ultrasound images will then be compared to the arthrogram findings, other imaging findings such as MRI and surgical pathological findings such as arthroscopy (if any.)
  Arms: Ultrasound Post-Arthrogram

SUMMARY:
The purpose of this study is to determine the usefulness of contrast in ultrasonography of the joints.

DETAILED DESCRIPTION:
To determine if using intra-articular contrast (contrast injected into a joint) will provide clearer, more precise ultrasound images of the joints then an ultrasound done without the use of a contrast agent.

ELIGIBILITY:
Inclusion Criteria:

* clinically ordered arthrogram

Exclusion Criteria:

* pregnant women
* children under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-09; Primary Completion 2010-08 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To add to the general knowledge of the researchers and to possibly benefit future patients in the diagnosis and treatment of joint abnormalities. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States